CLINICAL TRIAL: NCT01085435
Title: Evaluation oF Factors ImpacTing CLinical Outcome and Cost EffectiveneSS of the S-ICD (The EFFORTLESS S-ICD Registry)
Brief Title: Boston Scientific Post Market Subcutaneous-Implantable Cardioverter Defibrillator (S-ICD) Registry
Acronym: EFFORTLESS
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90904925; 90904928
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-11

CONDITIONS: Tachycardia, Ventricular
Keywords: ICD; defibrillator
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- EFFORTLESS Main Study: Patients implanted with a CE marked S-ICD System, not participating in Cameron Health's Investigational Device Exemption (IDE) Clinical Study.
  Interventions: Device: S-ICD System
- Extension Phase Sub Study: The Sub-Study patients were preferably recruited from the active EFFORTLESS S-ICD patient population. Patients, who had already completed the EFFORTLESS S-ICD Registry in the past, were considered secondarily for participation in the Sub-Study.
  Interventions: Device: S-ICD System

INTERVENTIONS:
Device: S-ICD System — The S-ICD System is an implantable technology that uses a subcutaneous pulse generator and subcutaneous electrode system to treat ventricular tachyarrhythmias. The S-ICD System consists of the pulse generator, subcutaneous electrode, the programmer and electrode insertion tool.
  Other Names: S-ICD Pulse Generator; S-ICD Subcutaneous Electrode; S-ICD Electrode Insertion Tool; S-ICD Programmer

SUMMARY:
The EFFORTLESS ICD Registry is an observational, standard of care evaluation designed to demonstrate the early, mid and long-term clinical effectiveness the Boston Scientific S-ICD System. In addition, analysis of resource utilization and costs will be performed to document treatment costs for periods defined by Registry endpoints. Protocol 90904928 restricts enrolment to patients over 18 years of age while protocol 90904925 allows all patients to be included.

DETAILED DESCRIPTION:
EFFORTLESS is an observational, post market, standard of care, Registry to be conducted at approximately 50 centers worldwide in patients requiring an ICD for the treatment of ventricular tachyarrhythmias. Patients included in the registry will have been implanted with the S-ICD system since its CE mark (commercial regulatory approval) and will be followed for up to 60 months. The patients' perception of their therapy will be evaluated using Quality of Life assessments and the Registry will include an exploratory analysis of resource utilization and costs based on measures of clinical outcome such as complication rates, unscheduled hospitalizations and length of stay. The objective will be to enable comparison of costs of the S-ICD system versus a standard transvenous system.

An Extension Phase Sub-Study will extend the EFFORTLESS S-ICD Registry in order to achieve an average of approximately 8 years of follow-up from index procedure. A subgroup of approximately 200 patients will be enrolled at a sub-set of EFFORTLESS sites. The data analysis will focus on long-term S-ICD system-related adverse events, S-ICD replacements and device longevity.

ELIGIBILITY:
Main study:

Inclusion Criteria

1. Age >/= 18yrs
2. Eligible for implantation of an S-ICD system per local clinical guidelines or currently implanted with an S-ICD system (Software (SW) version 1.59.0 or later)
3. Willing and able to provide written informed consent or have informed consent as provided by a legal representative

Exclusion Criteria:

1. Participation in any other investigational study that may interfere with interpretation of the Registry results
2. Incessant ventricular tachycardia and/or spontaneous, frequently recurring ventricular tachycardia that is reliably terminated with anti-tachycardia pacing
3. Patients with unipolar pacemakers or implanted devices that revert to unipolar pacing

Extension Phase Sub-study:

Inclusion Criteria

1. Subjects who are actively enrolled in the EFFORTLESS S-ICD Registry OR Subjects who completed the 5-year follow-up in the EFFORTLESS S-ICD Registry. All clinical events, spontaneous and induced episode data and system replacement or revision data since the last EFFORTLESS S-ICD Annual Follow-Up of the main study must be available in medical files or equivalent.
2. Subjects who are actively implanted with an S-ICD pulse generator (SQ-RX, EMBLEM or EMBLEM MRI) and an S-ICD electrode (Q-TRAK or EMBLEM) or any other future commercial available versions
3. Willing and able to provide written informed consent or have informed consent as provided by a legal representative and willing to participate in all testing and follow-ups as described the Sub-Study protocol
4. Age 18 or above, and of legal age to give informed consent specific to national laws

Exclusion Criteria

1. Subjects with device replacement from the S-ICD to a transvenous ICD
2. Subjects with unipolar pacemakers or implanted devices that revert to unipolar pacing
3. Subjects that are participating in any other investigational study that may interfere with interpretation of the Registry results, without the written approval of Boston Scientific

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post CE mark ICD patients eligible for implantation of the S-ICD system
Sampling Method: Non-Probability Sample
Enrollment: 994 (Actual)
Dates: Start 2011-02-02 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2024-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pier Lambiase, Prof., Study Chair — St. Bartholomew's Hospital, London
Locations (44):
- Na Homolce Hospital, Prague, Prague 5, Czechia
- Denmark (4):
  - Rigshospitalet, Copenhagen, København
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
- France (3):
  - CHU La Timone, Marseille
  - Nouvelles Cliniques Nantaises, Nantes
  - Hôpital Cardiologique du Haut-L'évêque, Pessac
- Germany (9):
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - Immanuel Klinikum Bernau Herzzentrum Brandenburg, Bernau
  - Klinikum Bielefeld, Bielefeld
  - Medizinische Hochschule Hannover, Hanover
  - University Hospital Schleswig-Holstein, Lübeck
  - Universitätsmedizin Mannheim, Mannheim
  - Ludwig-Maximilians-Universität München, Campus Großhadern, Munich
  - Universitätsklinikum Münster, Münster
  - Marienkrankenhaus Papenburg, Papenburg
- Italy (5):
  - Arnas Garibaldi Nesima, Catania
  - Ospedale Sacro Cuore Don Calabria, Negrar
  - Azienda Ospedaliero Universitaria Padova, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Policlinico Casilino, Rome
- Netherlands (7):
  - Maastricht University Medical Center, Maastricht, AZ Maastricht
  - Catharina Eindhoven Hospital, Eindhoven, EJ Eindhoven
  - Amsterdam Medisch Centrum, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - St Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medical Center, Rotterdam
- Auckland City Hospital, Auckland, New Zealand
- Hospital Santa Cruz, Carnaxide, Portugal
- Complexo Hospitalario Universitario, A Coruña, Spain
- United Kingdom (12):
  - Papworth Hospital, Cambridge, Cambridgeshire
  - Leeds General Infirmary, Leeds, Yorkshire
  - Royal Sussex County Hospital, Brighton
  - Bristol Royal Infirmary, Bristol
  - Russells Hall Hospital, Dudley
  - Yorkhill Children's Hospital, Glasgow
  - Yorkshire Heart Centre, Leeds
  - St. Bartholomew's Hospital, London
  - Kings College Hospital, London
  - John Radcliffe Hospital, Oxford
  - Northern General Hospital, Sheffield
  - Southampton General, Southampton

REFERENCES:
- [Derived] Boersma L, Barr C, Knops R, Theuns D, Eckardt L, Neuzil P, Scholten M, Hood M, Kuschyk J, Jones P, Duffy E, Husby M, Stein K, Lambiase PD; EFFORTLESS Investigator Group. Implant and Midterm Outcomes of the Subcutaneous Implantable Cardioverter-Defibrillator Registry: The EFFORTLESS Study. J Am Coll Cardiol. 2017 Aug 15;70(7):830-841. doi: 10.1016/j.jacc.2017.06.040. PMID 28797351
- [Derived] Burke MC, Gold MR, Knight BP, Barr CS, Theuns DAMJ, Boersma LVA, Knops RE, Weiss R, Leon AR, Herre JM, Husby M, Stein KM, Lambiase PD. Safety and Efficacy of the Totally Subcutaneous Implantable Defibrillator: 2-Year Results From a Pooled Analysis of the IDE Study and EFFORTLESS Registry. J Am Coll Cardiol. 2015 Apr 28;65(16):1605-1615. doi: 10.1016/j.jacc.2015.02.047. PMID 25908064
- [Derived] Lambiase PD, Barr C, Theuns DA, Knops R, Neuzil P, Johansen JB, Hood M, Pedersen S, Kaab S, Murgatroyd F, Reeve HL, Carter N, Boersma L; EFFORTLESS Investigators. Worldwide experience with a totally subcutaneous implantable defibrillator: early results from the EFFORTLESS S-ICD Registry. Eur Heart J. 2014 Jul 1;35(25):1657-65. doi: 10.1093/eurheartj/ehu112. Epub 2014 Mar 26. PMID 24670710

RESULTS

PARTICIPANT FLOW:
Period: Main Study
Arm/Group | EFFORTLESS Main Study
Started (signed consent) | 994
Baseline (implanted & followed) | 984
Completed | 703
Not Completed | 291
Period: EFFORTLESS Extension Phase Substudy
Arm/Group | EFFORTLESS Main Study
Started | 203
Completed | 164
Not Completed | 39

BASELINE CHARACTERISTICS:
Population: Patients implanted with a CE marked S-ICD System, not participating in Cameron Health's Investigational Device Exemption (IDE) Clinical Study.
  S-ICD System: The S-ICD System is an implantable technology that uses a subcutaneous pulse generator and subcutaneous electrode system to treat ventricular tachyarrhythmias. The S-ICD System consists of the pulse generator, subcutaneous electrode, the programmer and electrode insertion tool.
  Main Study
Arm/Group | EFFORTLESS Main Study
Number analyzed (Participants) | 984
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275
  Male | 709
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Perioperative S-ICD Complication Free Rate
Description: The number of subjects without Type I Complications within 30 Days of Implant divided by the Total Implanted Subjects.
Time Frame: 30 days post implant
Population: All implanted patients (N=984)
Measure: Count of Participants; unit: Participants
Arm/Group | EFFORTLESS Main Study
Number analyzed (Participants) | 984
Participants | 983

2. Primary Outcome: 360 Day S-ICD Complication Free Rate
Description: The Kaplan-Meier (KM) Survival Estimate of 360-Day Type I Complications.
Time Frame: Minimum 360 days post implant
Population: All implanted patients (N=984)
Measure: Count of Participants; unit: Participants
Arm/Group | EFFORTLESS Main Study
Number analyzed (Participants) | 984
Participants | 970

3. Primary Outcome: Percentage of Inappropriate Shocks for Atrial Fibrillation (AF)/Supraventricular Tachycardia (SVT)
Description: The number of subjects who received at least one inappropriate shock for SVT above the discrimination zone and SVT discriminator errors divided by the total implanted subjects.
Time Frame: From enrollment to 5-year annual visit.
Population: All implanted patients (N=984)
Measure: Count of Participants; unit: Participants
Arm/Group | EFFORTLESS Main Study
Number analyzed (Participants) | 984
Participants | 29

4. Other Pre Specified Outcome: Extension Phase Rate of Long-term S-ICD System-related Adverse Events
Description: Rate of adverse events related to the S-ICD system in subjects of the EFFORTLESS Extension Phase sub study
Time Frame: From enrollment in the Extension Phase up to 5 years until the 5th annual follow-up of the substudy, usually up to 60 months +/- 90 days.
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Number (95% Confidence Interval); unit: Percentage of Survival w/o l-term AE
Groups:
- Extension Phase Sub Study: Subset of Subjects, who had already completed the EFFORTLESS S-ICD Registry
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Percentage of Survival w/o l-term AE
  240 Days Post Replacement Procedure | 95.0 [92.1 to 98.0]
  360 Days Post Replacement Procedure | 94.6 [91.4 to 97.7]
  720 Days Post Replacement Procedure | 93.6 [90.2 to 96.9]
  1080 Days Post Replacement Procedure | 92.6 [88.9 to 96.2]
  1440 Days Post Replacement Procedure | 92.0 [88.3 to 95.8]
  1800 Days Post Replacement Procedure | 90.5 [86.2 to 94.8]
  2160 Days Post Replacement Procedure | 89.3 [84.6 to 94.0]

5. Other Pre Specified Outcome: Extension Phase S-ICD Replacements for Functionality
Description: Number of S-ICD replacements with another type of implantable defibrillator for functionality unavailable with an S-ICD, such as a need for additional brady therapy, cardiac resynchronization therapy, antitachycardia pacing, or other similar reasons
Time Frame: From enrollment into the Extension Phase up to 5 years until the 5th annual follow-up of the substudy, usually up to 60 months +/- 90 days.
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Number; unit: Subjects w. repl. for functionality
Units Other Than Participants: S-ICD replacements for functionality
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Number analyzed (S-ICD replacements for functionality) | 26
Subjects w. repl. for functionality
  Battery: Early Battery Depletion | 12
  Inappropriate Shocks | 5
  Change in Indication: Need Bi-V Pacing | 3
  Change in Indication: Need Additional ICD Programmability for VT | 1
  Change in Indication: Need Bradycardia Pacing | 1
  Investigator Discretion | 1
  MRI Compatibility | 1
  S-ICD PG Suspected Malfunction | 1
  Unknown reason for out of service | 1

6. Other Pre Specified Outcome: Extension Phase Device Longevity
Description: Minimum Implant Time (Days). The data includes information on devices tracked from the date of implant until they went out of service, as well as devices tracked from implant until the last available follow-up before the subject exited the study for any reason (such as study conclusion, death, or withdrawal). Devices still functioning at the end of their observation period continue to add to their longevity beyond this period. Thus, the reported value underestimates actual device longevity, representing only the minimum duration these devices were known to function.
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Mean (Standard Deviation); unit: Minimum Implant time [days]
Units Other Than Participants: pulse generators
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Number analyzed (pulse generators) | 418
Minimum Implant time [days]
  PG Model 1010: number analyzed (pulse generators) | 209
  PG Model 1010 | 2063.7 (494.1)
  PG Model A209: number analyzed (pulse generators) | 19
  PG Model A209 | 1539.1 (676.6)
  PG Model A219: number analyzed (pulse generators) | 190
  PG Model A219 | 1485.5 (630.3)

7. Other Pre Specified Outcome: Extension Phase Rate of Complications Related to the S-ICD Replacements
Description: K-M Estimate (%) for freedom of complications related to the S-ICD replacements
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Number (95% Confidence Interval); unit: percentage of freedom from complications
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
percentage of freedom from complications
  240 Days Post Replacement Procedure | 92.1 [88.4 to 95.8]
  360 Days Post Replacement Procedure | 91.1 [87.2 to 95.0]
  720 Days Post Replacement Procedure | 87.1 [82.5 to 91.7]
  1080 Days Post Replacement Procedure | 83.6 [78.5 to 88.7]
  1440 Days Post Replacement Procedure | 79.6 [74.0 to 85.2]
  1800 Days Post Replacement Procedure | 77.0 [70.9 to 83.1]
  2160 Days Post Replacement Procedure | 77.0 [70.6 to 83.4]

8. Other Pre Specified Outcome: Extension Phase Appropriate Shock Therapy for VT/VF
Description: K-M Estimate (%) for Freedom of appropriate shock therapy for VT/VF
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Number (95% Confidence Interval); unit: percentage of freedom of appr. shocks
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
percentage of freedom of appr. shocks
  240 Days Post Implant | 98.5 [96.8 to 100.0]
  360 Days Post Implant | 98.0 [96.1 to 99.9]
  720 Days Post Implant | 96.0 [93.3 to 98.7]
  1080 Days Post Implant | 94.0 [90.6 to 97.3]
  1440 Days Post Implant | 91.4 [87.2 to 95.5]
  1800 Days Post Implant | 85.4 [79.9 to 90.8]

9. Other Pre Specified Outcome: Extension Phase Inappropriate Shock Therapy
Description: K-M Estimate (%) for Freedom of Inappropriate Shock Therapy
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Number (95% Confidence Interval); unit: % of freedom of inappropriate shocks
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
% of freedom of inappropriate shocks
  240 Days Post Implant | 98.0 [96.1 to 99.9]
  360 Days Post Implant | 96.0 [93.3 to 98.7]
  720 Days Post Implant | 93.5 [90.1 to 96.9]
  1080 Days Post Implant | 90.0 [85.9 to 94.2]
  1440 Days Post Implant | 89.0 [84.6 to 93.4]
  1800 Days Post Implant | 88.0 [83.2 to 92.7]
  2160 Days Post Implant | 86.2 [80.9 to 91.5]

10. Other Pre Specified Outcome: Extension Phase VF Induction Testing at Replacement
Description: Percentage of VF induction testing at replacement
Time Frame: as for outcome 4
Population: Subjects participating in the Extension Phase for whom which VF induction testing was performed during the replacement procedures (N=33)
Measure: Count of Participants; unit: Participants
Groups:
- Ext. Phase Subjects for Whom VF Induction Testing Was Performed During the Replacement Procedures: Subjects participating in the Extension Phase for whom VF induction testing was performed during the replacement procedures (N=33)
Arm/Group | Ext. Phase Subjects for Whom VF Induction Testing Was Performed During the Replacement Procedures
Number analyzed (Participants) | 33
Participants
  Subjects with at least one evaluable conversion test: number analyzed (Participants) | 29
  Subjects with at least one evaluable conversion test: At least one Successful Conversion <= 65J | 27
  Subjects with at least one evaluable conversion test: Successful Conversions > 65J only | 1
  Subjects with at least one evaluable conversion test: Subjects with Successful Shock Energy NOT Documented | 1
  Subjects with at least one evaluable conversion test: All Conversions have Incomplete Data | 0
  Subjects with only non-evaluable conversion tests: number analyzed (Participants) | 4
  Subjects with only non-evaluable conversion tests: At least one Successful Conversion <= 65J | 0
  Subjects with only non-evaluable conversion tests: Successful Conversions > 65J only | 0
  Subjects with only non-evaluable conversion tests: Subjects with Successful Shock Energy NOT Documented | 0
  Subjects with only non-evaluable conversion tests: All Conversions have Incomplete Data | 4

11. Other Pre Specified Outcome: Extension Phase Additional Invasive Interventions
Description: Number of Additional invasive interventions
Time Frame: as for outcome 4
Measure: Number; unit: Number of Interventions
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Number of Interventions
  PG Revision | 13
  Electrode Revision | 5
  Major Cardiac Surgery Revision | 5
  Other, incl. blood draw, IV Rx, angio, cardioversion, PCI, ablation | 64

12. Other Pre Specified Outcome: Extension Phase Additional Invasive Interventions
Description: Number of subjects with additional invasive interventions
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Number; unit: participants w. add. inv. intervention
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
participants w. add. inv. intervention
  PG Revision | 13
  Electrode Revision | 5
  Major Cardiac Surgery Revision | 5
  Other, incl. blood draw, IV Rx, angio, cardioversion, PCI, ablation | 36

13. Other Pre Specified Outcome: Extension Phase Use of Anti-arrhythmic Drugs
Description: Number of subjects in the Extension Phase using anti-arrhythmic drugs
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Participants
  Class I - Sodium Channel Blockers: Disopyramide | 2
  Class I - Sodium Channel Blockers: Flecainide | 2
  Class I - Sodium Channel Blockers: Mexiletine | 2
  Class I - Sodium Channel Blockers: Quinidine | 1
  Class II - Beta Blockers: Atenolol | 5
  Class II - Beta Blockers: Bisoprolol | 79
  Class II - Beta Blockers: Carvedilol | 12
  Class II - Beta Blockers: Celiprolol | 1
  Class II - Beta Blockers: Metoprolol | 34
  Class II - Beta Blockers: Nadolol | 1
  Class II - Beta Blockers: Nebivolol | 7
  Class II - Beta Blockers: Propranolol | 2
  Class III - Potassium Channel Blockers: Amiodarone | 24
  Class III - Potassium Channel Blockers: Sotalol | 8
  Class IV - Calcium Channel Blockers: Amlodipine | 5
  Class IV - Calcium Channel Blockers: Diltiazem | 3
  Class IV - Calcium Channel Blockers: Felodipine | 1
  Class IV - Calcium Channel Blockers: Verapamil | 8

14. Other Pre Specified Outcome: Extension Phase Ventricular Rate of Episodes (Mean)
Description: Ventricular rate in of episodes in beats per minute
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Mean (Standard Deviation); unit: episodes
Units Other Than Participants: episodes
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Number analyzed (episodes) | 60
episodes
  Rate of observed discrete MVT Episodes: number analyzed (episodes) | 34
  Rate of observed discrete MVT Episodes | 217.5 (33.3)
  Rate of observed discrete PVT/VF Episodes: number analyzed (episodes) | 26
  Rate of observed discrete PVT/VF Episodes | 269.6 (51.1)

15. Other Pre Specified Outcome: Extension Phase Ventricular Rate of Episodes (Median)
Description: Ventricular rate in of episodes in beats per minute
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Median (Full Range); unit: beats per minute
Units Other Than Participants: episodes
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Number analyzed (episodes) | 60
beats per minute
  Rate of observed discrete MVT Episodes: number analyzed (episodes) | 34
  Rate of observed discrete MVT Episodes | 210 [120 to 320]
  Rate of observed discrete PVT/VF Episodes: number analyzed (episodes) | 26
  Rate of observed discrete PVT/VF Episodes | 260 [200 to 400]

16. Other Pre Specified Outcome: Extension Phase Ventricular Rate of Episodes (IQR)
Description: Ventricular rate in of episodes in beats per minute
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Mean (Inter-Quartile Range); unit: beats per minute
Units Other Than Participants: episodes
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Number analyzed (episodes) | 60
beats per minute
  Rate of observed discrete MVT Episodes: number analyzed (episodes) | 34
  Rate of observed discrete MVT Episodes | 217.5 [200 to 240]
  Rate of observed discrete PVT/VF Episodes: number analyzed (episodes) | 26
  Rate of observed discrete PVT/VF Episodes | 269.6 [240 to 300]

17. Other Pre Specified Outcome: Extension Phase Ventricular Rate of Non-Sustained Episodes (Mean)
Description: Ventricular rate in of episodes in beats per minute
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Mean (Standard Deviation); unit: beats per minute
Units Other Than Participants: episodes
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Number analyzed (episodes) | 83
beats per minute
  Rate of observed Non-Sustained MVT Episodes: number analyzed (episodes) | 73
  Rate of observed Non-Sustained MVT Episodes | 212.3 (25.8)
  Rate of observed Non-Sustained PVT/VF Episodes: number analyzed (episodes) | 10
  Rate of observed Non-Sustained PVT/VF Episodes | 248.4 (60.0)

18. Other Pre Specified Outcome: Extension Phase Ventricular Rate of Non-Sustained Episodes (Median)
Description: Ventricular rate in of episodes in beats per minute
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Median (Full Range); unit: beats per minute
Units Other Than Participants: episodes
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Number analyzed (episodes) | 83
beats per minute
  Rate of observed Non-Sustained MVT Episodes: number analyzed (episodes) | 73
  Rate of observed Non-Sustained MVT Episodes | 200 [180 to 300]
  Rate of observed Non-Sustained PVT/VF Episodes: number analyzed (episodes) | 10
  Rate of observed Non-Sustained PVT/VF Episodes | 245 [184 to 400]

19. Other Pre Specified Outcome: Extension Phase Ventricular Rate of Non-Sustained Episodes (IQR)
Description: Ventricular rate in of episodes in beats per minute
Time Frame: as for outcome 4
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Mean (Inter-Quartile Range); unit: beats per minute
Units Other Than Participants: episodes
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Number analyzed (episodes) | 83
beats per minute
  Rate of observed Non-Sustained MVT Episodes: number analyzed (episodes) | 73
  Rate of observed Non-Sustained MVT Episodes | 212.3 [200 to 220]
  Rate of observed Non-Sustained PVT/VF Episodes: number analyzed (episodes) | 10
  Rate of observed Non-Sustained PVT/VF Episodes | 248.4 [210 to 260]

20. Other Pre Specified Outcome: Complication Events
Description: Summary of all reported complications defined as a clinical event that results in invasive intervention.
Time Frame: From enrollment in the initial main study until the 5th annual follow-up of the substudy.
Population: All subjects enrolled in the EFFORTLESS Extension Phase Sub Study (N=203)
Measure: Count of Units; unit: events
Units Other Than Participants: events
Arm/Group | Extension Phase Sub Study
Number analyzed (Participants) | 203
Number analyzed (events) | 105
events
  Abnormal Thyroid Condition | 1
  Adverse Reaction (Medications) (Non-System/Non-Procedure related) | 1
  Adverse Reaction (Respiratory) | 1
  Anemia | 1
  Atrial Fibrillation/Flutter (Cardiac) | 6
  Cancer | 3
  Cardiac Arrest | 4
  Chest Pain (Cardiac) | 1
  Coronary Artery Disease | 6
  Death (as stand-alone event) | 2
  Electrode Movement | 1
  Erosion | 2
  Fracture/Broken Bone | 2
  GI Disorder | 2
  HEENT Disorder | 1
  Heart Failure/Worsening of Heart Failure | 17
  Hematoma not related to TV-ICD Placement | 2
  Hematoma related to TV-ICD Placement | 1
  Inappropriate Shock: Cardiac Oversensing | 3
  Inappropriate Shock: Non-Cardiac Oversensing | 2
  Inappropriate Shock: SVT Above Discrimination Zone (Normal Device Function) | 1
  Infection not related to S-ICD System | 3
  Inflammation (Non-Cardiac/Non-System/Non-Procedure related) | 1
  Multi-system Failure | 2
  Other (Non-Cardiac/Non-System/Non-Procedure related) | 1
  Other: Cardiac (Non-System/Procedure related) | 1
  Pain/Discomfort (Non-Cardiac/Non-System/Non-Procedure related) | 2
  Peripheral Vascular Disease | 1
  Pneumonia | 4
  Premature Cell Battery Depletion: Premature Declaration | 5
  Premature Cell Battery Depletion: Random Component Failure | 2
  Respiratory Failure (Non-Cardiac/Non-System/Non-Procedure related) | 1
  Shortness of Breath, Dyspnea (Non-Cardiac/Non-System/Non-Procedure related) | 1
  Skeletal/ Muscular Injury | 1
  Syncope (Non-Cardiac/Non-System/Non-Procedure related) | 2
  System Infection | 1
  Unable to Convert: During Procedure | 1
  Worsening of Benign Prostatic Hyperplasia | 1
  Worsening of VT/VF | 15

ADVERSE EVENTS:
Time Frame: From enrollment to 5-year annual visit.
Arm/Group | EFFORTLESS Main Study
All-Cause Mortality (participants affected / at risk) | 91/984
Serious Adverse Events (participants affected / at risk) | 199/984
Other Adverse Events (participants affected / at risk) | 531/984
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EFFORTLESS Main Study (N=984)
Inappropriate Shock: SVT Above Discrimination Zone (Normal Device Function) (Product Issues) | 1 (1)
Inappropriate Shock: Cardiac Oversensing (Product Issues) | 10 (11)
Inappropriate Shock: Non-Cardiac Oversensing (Product Issues) | 1 (1)
PG Movement (Product Issues) | 2 (2)
Erosion (Product Issues) | 3 (3)
Inability to Communicate with the Device (Product Issues) | 1 (1)
Fear of Shocks (Psychiatric disorders) | 1 (1)
Imminent Erosion (Product Issues) | 1 (1)
Suspected Device Malfunction (Product Issues) | 1 (1)
Incision/Superficial Infection (Infections and infestations) | 1 (1)
System Infection (Infections and infestations) | 9 (9)
Atrial Fibrillation/Flutter (Procedure related) (Cardiac disorders) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Sub-optimal Electrode position (Injury, poisoning and procedural complications) | 1 (1)
Adverse Reaction (Medications) (Injury, poisoning and procedural complications) | 1 (1)
Adverse Reaction (General) (Injury, poisoning and procedural complications) | 1 (1)
Electrode Movement (Product Issues) | 1 (1)
Bleeding (Procedure related) (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Limited Emphysema (Injury, poisoning and procedural complications) | 1 (1)
Atrial Fibrillation/Flutter (Cardiac) (Cardiac disorders) | 7 (9)
Heart Failure/Worsening of Heart Failure (Cardiac disorders) | 46 (53)
Myocardial Infarction (Cardiac disorders) | 8 (8)
Cardiac Arrest (Cardiac disorders) | 3 (3)
Thrombosis (Blood and lymphatic system disorders) | 2 (3)
Syncope (Cardiac) (Cardiac disorders) | 3 (3)
Worsening of VT/VF (Cardiac disorders) | 15 (18)
Coronary Artery Disease (Cardiac disorders) | 10 (10)
Angina (Cardiac disorders) | 1 (1)
Chest Pain (Cardiac) (Cardiac disorders) | 1 (1)
Peripheral Vascular Disease (Vascular disorders) | 6 (6)
Bradycardia/AV Block (Cardiac disorders) | 3 (3)
Right Bundle Branch Block (Cardiac disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Stroke (Non-System/Non-Procedure related) (Vascular disorders) | 7 (7)
Infection not related to S-ICD System (Infections and infestations) | 16 (17)
Psychological Disorder (Psychiatric disorders) | 3 (4)
Pain/Discomfort (Non-Cardiac/Non-System/Non-Procedure related) (General disorders) | 1 (1)
Pneumothorax (Non-System/Non-Procedure related) (Injury, poisoning and procedural complications) | 1 (1)
GI Disorder (Gastrointestinal disorders) | 5 (5)
Abnormal Thyroid Condition (Endocrine disorders) | 2 (2)
Bleeding (Non-System/Non-Procedure related) (Injury, poisoning and procedural complications) | 7 (7)
Implant/Replacement of Any Concomitant Device (Product Issues) | 1 (1)
Fracture/Broken Bone (Injury, poisoning and procedural complications) | 4 (4)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11)
Kidney Disease (Renal and urinary disorders) | 8 (9)
Trauma (Non-Cardiac/Non-System/Non-Procedure related) (Injury, poisoning and procedural complications) | 3 (3)
HEENT Disorder (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Death (General disorders) | 7 (7) — Cause unknown, no information available to determine the cause of the death
Neurological (General disorders) | 1 (1)
Other (Non-Cardiac/Non-System/Non-Procedure related) (General disorders) | 2 (2)
Metabolic Disorder (Metabolism and nutrition disorders) | 3 (3)
Multi-system Failure (General disorders) | 18 (18)
Other: Cardiac (Non-System/Procedure related) (Cardiac disorders) | 2 (2)
Respiratory Failure (Non-Cardiac/Non-System/Non-Procedure related) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Unable to Convert: During Procedure (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EFFORTLESS Main Study (N=984)
Inappropriate Shock: SVT Above Discrimination Zone (Normal Device Function) (Product Issues) | 23 (35)
Inappr. Shock: Conv. bef. shock (Normal Function) (Product Issues) | 1 (1) — Inappropriate Shock: Ventricular Tachycardia (VT)/Ventricular Fibrillation (VF) spontaneously converted immediately before shock (Normal Device Function)
Inappropriate Shock: Cardiac Oversensing (Product Issues) | 105 (148)
Adverse Reaction (Bradycardia) (Injury, poisoning and procedural complications) | 2 (2)
Inappropriate Shock: Non-Cardiac Oversensing (Product Issues) | 25 (28)
Adverse Reaction (Medications) (Injury, poisoning and procedural complications) | 4 (4)
Inappropriate Shock: Discrimination Error (Product Issues) | 6 (7)
Adverse Reaction (Respiratory) (Injury, poisoning and procedural complications) | 1 (1)
Phantom Shock (Product Issues) | 10 (10)
Premature Cell Battery Depletion: Premature Declaration (Product Issues) | 3 (3)
Atrial Fibrillation/Flutter (Procedure related) (Cardiac disorders) | 5 (5)
Premature Cell Battery Depletion: Random Component Failure (Product Issues) | 5 (5)
Bleeding (Procedure related) (Injury, poisoning and procedural complications) | 2 (2)
PG Movement (Product Issues) | 8 (9)
Inability to Communicate with the Device (Product Issues) | 2 (2)
Phantom Vibration (Psychiatric disorders) | 1 (1)
Phantom Beeps (Psychiatric disorders) | 1 (1)
Erosion (Product Issues) | 16 (16)
Discomfort (Product Issues) | 74 (87)
Imminent Erosion (Product Issues) | 4 (4)
Electrode Movement (Product Issues) | 8 (8)
Fear of Shocks (Psychiatric disorders) | 11 (12)
Electrode damaged and replaced during concomitant device procedure (Product Issues) | 1 (1)
Suspected Device Malfunction (Product Issues) | 1 (1)
Undersensing: Defibrillation (Product Issues) | 1 (1)
Fever (Infections and infestations) | 3 (3)
Fluid Accumulation (Procedure related) (Injury, poisoning and procedural complications) | 1 (1)
Programmer/Software Error code (Product Issues) | 1 (1)
Inappropriate Post Shock Pacing (Product Issues) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 30 (34)
Inadequate Pocket Size (Injury, poisoning and procedural complications) | 1 (1)
Inadequate/Prolonged Healing of Incision Site (Injury, poisoning and procedural complications) | 8 (8)
Incision/Superficial Infection (Infections and infestations) | 24 (24)
Keloid (Skin and subcutaneous tissue disorders) | 1 (1)
Nerve Damage (Procedure related) (Injury, poisoning and procedural complications) | 3 (3)
System Infection (Infections and infestations) | 24 (26)
Sub-optimal Electrode position (Injury, poisoning and procedural complications) | 7 (7)
Syncope (Procedure related) (Injury, poisoning and procedural complications) | 1 (1)
Sub-optimal PG position (Injury, poisoning and procedural complications) | 1 (1)
Sub-optimal PG and Electrode position (Injury, poisoning and procedural complications) | 3 (3)
Redness/Irritation (Injury, poisoning and procedural complications) | 13 (14)
Seroma (Injury, poisoning and procedural complications) | 4 (4)
Subcutaneous Emphysema (Injury, poisoning and procedural complications) | 1 (1)
Suture Discomfort (Product Issues) | 6 (6)
Device Malfunction (Product Issues) | 1 (1)
Other (Procedure related: PG) (Product Issues) | 2 (2)
Other (Procedure related: Electrode) (Product Issues) | 1 (1)
Atrial Fibrillation/Flutter (Cardiac) (Cardiac disorders) | 34 (74)
Heart Failure/Worsening of Heart Failure (Cardiac disorders) | 48 (87)
Hypotension (Vascular disorders) | 3 (3)
Myocardial Infarction (Cardiac disorders) | 8 (8)
Thrombosis (Blood and lymphatic system disorders) | 6 (7)
Syncope (Cardiac) (Cardiac disorders) | 22 (27)
Near Syncope/Dizziness/Shortness of Breath/Confusion (Cardiac) (Cardiac disorders) | 19 (21)
VT below Conditional Zone (Cardiac disorders) | 3 (3)
Worsening of VT/VF (Cardiac disorders) | 69 (105)
Palpitations (Cardiac disorders) | 34 (42)
Coronary Artery Disease (Cardiac disorders) | 7 (8)
Chest Pain (Cardiac) (Cardiac disorders) | 24 (28)
Peripheral Vascular Disease (Vascular disorders) | 6 (6)
Bradycardia/AV Block (Cardiac disorders) | 14 (14)
Inflammation (Cardiac) (Infections and infestations) | 2 (2)
Right Bundle Branch Block (Cardiac disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Stroke (Non-System/Non-Procedure related) (Vascular disorders) | 5 (5)
Syncope (Non-Cardiac/Non-System/Non-Procedure related) (Cardiac disorders) | 14 (15)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Infection not related to S-ICD System (Infections and infestations) | 24 (26)
Hematoma (Non-System/Non-Procedure related) (Injury, poisoning and procedural complications) | 4 (4)
Hematoma (Post Explant of S-ICD System) (Injury, poisoning and procedural complications) | 1 (1)
Near Syncope/Dizziness/Shortness of Breath/Confusion (Non-Cardiac/Non-System/Non-Procedure related) (Cardiac disorders) | 18 (20)
Shortness of Breath, Dyspnea (Non-Cardiac/Non-System/Non-Procedure related) (Cardiac disorders) | 13 (13)
Psychological Disorder (Psychiatric disorders) | 13 (13)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pain/Discomfort (Non-Cardiac/Non-System/Non-Procedure related) (General disorders) | 21 (27)
Acute Appendicitis (Gastrointestinal disorders) | 1 (1)
Pleural Effusion (Non-System/Non-Procedure related) (Injury, poisoning and procedural complications) | 1 (2)
GI Disorder (Gastrointestinal disorders) | 27 (37)
Abnormal Thyroid Condition (Endocrine disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Bleeding (Non-System/Non-Procedure related) (Injury, poisoning and procedural complications) | 8 (10)
Nausea/Vomiting (General disorders) | 3 (3)
Repositioning of Any Concomitant Device (Product Issues) | 1 (1)
Implant/Replacement of Any Concomitant Device (Product Issues) | 7 (8)
Inflammation (Non-Cardiac/Non-System/Non-Procedure related) (Infections and infestations) | 7 (7)
Fracture/Broken Bone (Injury, poisoning and procedural complications) | 11 (12)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Kidney Disease (Renal and urinary disorders) | 12 (16)
Trauma (Non-Cardiac/Non-System/Non-Procedure related) (Injury, poisoning and procedural complications) | 9 (11)
HEENT Disorder (Respiratory, thoracic and mediastinal disorders) | 14 (18)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Fluid Accumulation (Non-Cardiac/Non-System/Non-Procedure related) (General disorders) | 1 (1)
Flu (General disorders) | 1 (1)
Genital/Urinary (General disorders) | 1 (1)
Neurological (General disorders) | 1 (1)
Other (Non-Cardiac/Non-System/Non-Procedure related) (General disorders) | 11 (11)
Metabolic Disorder (Metabolism and nutrition disorders) | 5 (6)
Abnormal Lab Values (Cardiac disorders) | 1 (1)
Mitral Insufficiency (Cardiac disorders) | 1 (1)
Other: Cardiac (Non-System/Procedure related) (Cardiac disorders) | 9 (9)
Respiratory Failure (Non-Cardiac/Non-System/Non-Procedure related) (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Unable to Convert: During Procedure (General disorders) | 9 (9)
Adverse Reaction (Medications) (Non-System/Non-Procedure related) (General disorders) | 2 (2)
Altered Mental Status (Psychiatric disorders) | 1 (1)
Hypertension (General disorders) | 3 (3)
Muscle Stimulation (Non-System/Non-Procedure related) (Injury, poisoning and procedural complications) | 2 (3)
SVT (Cardiac disorders) | 4 (4)
Unable to Convert: During Spontaneous Episode (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Consultant (PI) acknowledges and agrees that (i) Consultant shall not publish any data, report, white papers or other materials arising out of the Services performed pursuant to this Agreement without the prior written consent of Boston Scientific, and (ii) any such publication shall not include Boston Scientific Confidential Information except prior written consent of Boston Scientific.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT01085435/Prot_SAP_000.pdf